CLINICAL TRIAL: NCT01587248
Title: Harmonic Scalpel vs. Electrocautery Dissection in Modified Radical Mastectomy: A Randomized Controlled Trial
Brief Title: Use of Harmonic in Breast Surgery
Acronym: HMRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ghulam Murtaza, Co Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1519-Sur-ERC-10
Record Dates: First submitted 2012-04-19; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer; Modified Radical Mastectomy
Keywords: Breast cancer,; Harmonic scalpel,; Electrocautery,; Modified Radical Mastectomy,; Randomized Controlled Trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Second Harmonic Generation Microscopy; Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrocautery (Active Comparator): Raising of the flaps with electrocautery
  Interventions: Procedure: electrocautery
- Harmonic (Experimental): Dissection with harmonic scalpel in modified radical mastectomy
  Interventions: Device: Harmonic

INTERVENTIONS:
Device: Harmonic — Dissection with harmonic scalpel
  Arms: Harmonic
Procedure: electrocautery — Dissection in modified radical mastectomy
  Arms: Electrocautery

SUMMARY:
To compare harmonic scalpel with electrocautery for outcomes i.e. estimated blood loss (EBL), operating time, drain Volume and drain Days, seroma formation, surgical site infection and postoperative pain in adult females undergoing MRM at a tertiary care hospital. We hypothesized that harmonic yields better outcome than electrocautery dissection.

DETAILED DESCRIPTION:
In this randomized controlled trial, adult females who underwent MRM between April 2010 and July 2011 were randomized to receive either intervention A (harmonic scalpel) or B (electrocautery). The procedure was standardized except elevation of flaps and axillary dissection, that was performed as per randomization. Patients were followed up in clinic for four weeks. The outcomes were estimated blood loss (EBL), operating time, drain Volume and drain Days, complications (seroma, surgical site infection, hematoma and flap necrosis) and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult females with biopsy proven breast cancer underwent MRM

Exclusion Criteria:

* Simultaneous procedure (Reconstruction, Sentinel lymph node biopsy)

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Duration of drains (days) | 30 days
  Durations of drains in place after MRM: Patients were followed in clinic every 3rd day and drains were removed once the volume was <30ml a day.

SECONDARY OUTCOMES:
Operative time | 3-4 hours
  Time taken in minutes from incision to skin closure
Drain Volume | 30 days
  Daily charting of drain volume at a specified time with regular recording in routine clinic follow ups till the drains were is place.
Overall complications | 30 days
  Patients were followed up till 3o days. If any of the following were found, the patient was labelled to have complication:
  Seroma- fluctuant swelling under the flaps; SSI- as per CDC criteria; Hematoma- swelling under flaps with characteristic bruising; Flap necrosis- partial or complete necrosis of flaps.
Pain | 24 hours
  Pain was measured by Visual Analogue score (1-10) by a registered nurse at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shaista M Khan, FRCS, Study Chair — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Khan S, Khan S, Chawla T, Murtaza G. Harmonic scalpel versus electrocautery dissection in modified radical mastectomy: a randomized controlled trial. Ann Surg Oncol. 2014 Mar;21(3):808-14. doi: 10.1245/s10434-013-3369-8. PMID 24232511